CLINICAL TRIAL: NCT01954953
Title: European Research Projects on Rare Diseases Driven by Young Investigators
Brief Title: Clinical and Genetic Examination of Usher Syndrome Patients' Cohort in Europe
Acronym: EURUSH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: P13-02
Record Dates: First submitted 2013-09-18; First posted 2013-10-07 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2013-09

CONDITIONS: Usher Syndrome
Keywords: Retinitis Pigmentosa Syndromic; Congenital Deafness; Usher Syndrome Retinitis Pigmentosa and Deafness; Progressive Hearing Loss; Retinitis Pigmentosa
MeSH Terms: conditions — Usher Syndromes; Deafness; Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- no intervention

SUMMARY:
This study aims to characterize Usher patients in order to correlate this data with genetic information.

Tasks:

* Standardization and improvement of Usher syndrome diagnosis: refine and elaborate special tests of visual and otological function in association with genotype that enable to determine the most significant markers for Usher disease progression and therapeutic effect.
* Perform genotype and phenotype correlations in Usher syndrome patients
* Develop and maintain database for phenotypically and genotypically well-characterized patient cohorts, suitable for future therapeutic trials

ELIGIBILITY:
Inclusion criteria :

* Clinical characteristics for USH1, USH2 and USH3 as defined by the Usher syndrome consortium;
* Informed consent and agreement to participate in the study;
* Distance best corrected visual acuity ≥ 0.1.

Exclusion criteria:

* Systemic pathologies or severe ocular pathologies, systemic or topical medication usage, and/or other otolaryngology pathologies which could contaminate the results;
* Unwillingness to provide a blood sample ;
* Unwilling and/or unable to undergo the study procedures.

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: USH1, USH2 and USH3 as defined by the Usher syndrome consortium
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Genotype and phenotype correlations in Usher syndrome patients | up to 3 years (2016)
  Protocol outline: patients undergo clinical and molecular studies. These include extensive ophthalmologic (best corrected visual acuity, refraction, tonometry, color vision, visual field testing, pupillography*, full-field electroretinogram, multifocal electroretinogram, autofluorescence imaging, optical coherence tomography, adaptive optics*) examination, audiologic and vestibular evaluation and obtaining blood samples for genetic analysis.
  *only if available

CONTACTS AND LOCATIONS:
Locations (6):
- France (2):
  - CHU, Laboratoire de génétique moléculaire, INSERM, Montpellier
  - CIC of CHNO des Quinze-vingts, Paris
- Johannes Gutenberg University of Mainz, Institute of Zoology, Dept. Cell and Matrix Biology Mainz, Mainz, Germany
- Radboud University Nijmegen Medical Centre, Dept. Otorhinolaryngology, Nijmegen, Netherlands
- Portugal (2):
  - AIBILI, 4C - Coimbra Coordinating Centre for Clinical Research, Coimbra
  - IBILI- Faculty of Medicine - University of Coimbra, Center for Hereditary Diseases and Visual Neurosciences Laboratory, Coimbra

REFERENCES:
- [Background] Sliesoraityte I, Troeger E, Bernd A, Kurtenbach A, Zrenner E. Correlation between spectral domain OCT retinal nerve fibre layer thickness and multifocal pattern electroretinogram in advanced retinitis pigmentosa. Adv Exp Med Biol. 2012;723:471-8. doi: 10.1007/978-1-4614-0631-0_59. No abstract available. PMID 22183366
- [Background] Overlack N, Goldmann T, Wolfrum U, Nagel-Wolfrum K. Gene repair of an Usher syndrome causing mutation by zinc-finger nuclease mediated homologous recombination. Invest Ophthalmol Vis Sci. 2012 Jun 26;53(7):4140-6. doi: 10.1167/iovs.12-9812. PMID 22661463
- [Background] Goldmann T, Rebibo-Sabbah A, Overlack N, Nudelman I, Belakhov V, Baasov T, Ben-Yosef T, Wolfrum U, Nagel-Wolfrum K. Beneficial read-through of a USH1C nonsense mutation by designed aminoglycoside NB30 in the retina. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6671-80. doi: 10.1167/iovs.10-5741. Epub 2010 Jul 29. PMID 20671281
- [Background] Kersten FF, van Wijk E, Hetterschijt L, Baubeta K, Peters TA, Aslanyan MG, van der Zwaag B, Wolfrum U, Keunen JE, Roepman R, Kremer H. The mitotic spindle protein SPAG5/Astrin connects to the Usher protein network postmitotically. Cilia. 2012 Apr 25;1(1):2. doi: 10.1186/2046-2530-1-2. PMID 23351521
- [Background] Overlack N, Kilic D, Bauss K, Marker T, Kremer H, van Wijk E, Wolfrum U. Direct interaction of the Usher syndrome 1G protein SANS and myomegalin in the retina. Biochim Biophys Acta. 2011 Oct;1813(10):1883-92. doi: 10.1016/j.bbamcr.2011.05.015. Epub 2011 Jul 13. PMID 21767579
- [Background] Estrada-Cuzcano A, Koenekoop RK, Senechal A, De Baere EB, de Ravel T, Banfi S, Kohl S, Ayuso C, Sharon D, Hoyng CB, Hamel CP, Leroy BP, Ziviello C, Lopez I, Bazinet A, Wissinger B, Sliesoraityte I, Avila-Fernandez A, Littink KW, Vingolo EM, Signorini S, Banin E, Mizrahi-Meissonnier L, Zrenner E, Kellner U, Collin RW, den Hollander AI, Cremers FP, Klevering BJ. BBS1 mutations in a wide spectrum of phenotypes ranging from nonsyndromic retinitis pigmentosa to Bardet-Biedl syndrome. Arch Ophthalmol. 2012 Nov;130(11):1425-32. doi: 10.1001/archophthalmol.2012.2434. PMID 23143442
- [Background] Garcia-Garcia G, Besnard T, Baux D, Vache C, Aller E, Malcolm S, Claustres M, Millan JM, Roux AF. The contribution of GPR98 and DFNB31 genes to a Spanish Usher syndrome type 2 cohort. Mol Vis. 2013;19:367-73. Epub 2013 Feb 13. PMID 23441107
- [Background] Vache C, Besnard T, le Berre P, Garcia-Garcia G, Baux D, Larrieu L, Abadie C, Blanchet C, Bolz HJ, Millan J, Hamel C, Malcolm S, Claustres M, Roux AF. Usher syndrome type 2 caused by activation of an USH2A pseudoexon: implications for diagnosis and therapy. Hum Mutat. 2012 Jan;33(1):104-8. doi: 10.1002/humu.21634. Epub 2011 Nov 16. PMID 22009552
- [Background] Stoetzel C, Laurier V, Davis EE, Muller J, Rix S, Badano JL, Leitch CC, Salem N, Chouery E, Corbani S, Jalk N, Vicaire S, Sarda P, Hamel C, Lacombe D, Holder M, Odent S, Holder S, Brooks AS, Elcioglu NH, Silva ED, Rossillion B, Sigaudy S, de Ravel TJ, Lewis RA, Leheup B, Verloes A, Amati-Bonneau P, Megarbane A, Poch O, Bonneau D, Beales PL, Mandel JL, Katsanis N, Dollfus H. BBS10 encodes a vertebrate-specific chaperonin-like protein and is a major BBS locus. Nat Genet. 2006 May;38(5):521-4. doi: 10.1038/ng1771. Epub 2006 Apr 2. PMID 16582908
- [Background] Castelo-Branco M, Mendes M, Sebastiao AR, Reis A, Soares M, Saraiva J, Bernardes R, Flores R, Perez-Jurado L, Silva E. Visual phenotype in Williams-Beuren syndrome challenges magnocellular theories explaining human neurodevelopmental visual cortical disorders. J Clin Invest. 2007 Dec;117(12):3720-9. doi: 10.1172/JCI32556. PMID 18037993
- [Background] Goldmann T, Overlack N, Wolfrum U, Nagel-Wolfrum K. PTC124-mediated translational readthrough of a nonsense mutation causing Usher syndrome type 1C. Hum Gene Ther. 2011 May;22(5):537-47. doi: 10.1089/hum.2010.067. Epub 2011 Mar 25. PMID 21235327
- See also: Institut de la Vision — http://www.institut-vision.org/index.php?lang=en